CLINICAL TRIAL: NCT03284671
Title: Transcranial Direct Current Stimulation to Treat Patients With Severe and Resistant Obsessive Compulsive Disorders -Pilot Study (tDCS-TOC Pilot)
Brief Title: tDCS Stimulation to Treat Patients With Severe and Resistant Obsessive Compulsive Disorder-Pilot Study
Acronym: tDCS-TOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tDCS-TOC pilote
Record Dates: First submitted 2017-09-07; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Obsessive-compulsive Disorders and Symptoms
Keywords: Transcranial Direct Current Stimulation; Supplementary motor area; Orbitofrontal cortex
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bifocal stimulation (Experimental): Transcranial direct current Bifocal stimulation
  Interventions: Other: bifocal stimulation with tDCS

INTERVENTIONS:
Other: bifocal stimulation with tDCS — Patients will receive an active Treatment with tDCS (10 sessions of 30 mn with an intensity of 2 mA)

SUMMARY:
The purpose is to show that bifocal tDCS with an anodal stimulation on the orbitofrontal cortex and cathodic stimulation on supplementary motor areas is an effective treatment for patients with resistant and severe obsessive compulsive disorders.

ELIGIBILITY:
Patients must present all of the following criteria in order to be eligible:

Inclusion Criteria:

* Meets criteria for obsessive compulsive disorder according to DSM-IV with a "good insight" (BABS),
* Age: Participants will be both males and females, 18-70 years of age included.
* No current depressive and suicidal risks,
* No epileptic pathology,
* Chronic evolution ( Total Y-BOCS>20 ),
* Obsessive compulsive disorder resistant to pharmacology treatment, at least 2 antidepressants (type IRS) or cognitive and comportment therapy since at least one year,
* Stability treatment (antidepressants) for more than 12 weeks without significant improvement,
* Affiliation to a social security system (recipient or assignee),
* Signed written inform consent form.

Exclusion Criteria:

* Female subject who is pregnant, or of child-bearing age, sexually active and not using reliable contraception or who is nursing,
* Patient under curators
* Meets another diagnosis of axe 1 of DSM-IV,
* Current depressive or suicidal risks,
* Patient with a benzodiazepine treatment,
* Patient with any form of metal in the cranium, a pacemaker, skull defects, or skin lesions to the scalp (cuts, abrasions, rash) ,
* Epileptic patient,
* Patient with a medical history of cranial trauma,
* Patient unable to give his or hers informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2016-02-19 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is used to show that bifocal tDCS with anodal stimulation on OFC and cathodic stimulation on the SMA is an effective treatment | Day 14
  Score improvement on the Y-BOCS after 14 days compared to the baseline

SECONDARY OUTCOMES:
Evaluate the persistence of therapeutic response at 45 days | Day 45
  Score improvement on the Y-BOCS after 45 days compared to the baseline
Evaluate the persistence of therapeutic response at 105 days | Day 105
  Score improvement on the Y-BOCS after 105 days compared to the baseline
Evaluate the therapeutic effect of tDCS on the depressive and anxious symptoms associated with Obsessive compulsive disorder at 14 days | Day 14
  Score improvement of Hamilton and HDRS scales between the baseline and day 14
Evaluate the therapeutic effect of tDCS on the depressive and anxious symptoms associated with Obsessive compulsive disorder at 45 days | Day 45
  Score improvement of Hamilton and HDRS scales between the baseline and day 45
Evaluate the therapeutic effect of tDCS on the depressive and anxious symptoms associated with Obsessive compulsive disorder at 105 days | Day 105
  Score improvement of Hamilton and HDRS scales between the baseline and day 105
Evaluate the effect of tDCS on the quality of life at day 14 | Day 14
  Improvement of MOS SF-36 scale (Medical Outcome Study, Short Form) between baseline and day 14
Evaluate the effect of tDCS on the quality of life at day 45 | Day 45
  Improvement of MOS SF-36 scale (Medical Outcome Study, Short Form) between baseline and day 45
Evaluate the effect of tDCS on global functioning at day 14 | Day 14
  Improvement of GAF (Global Assessment of Functioning) scale between baseline and day 14
Evaluate the effect of tDCS on global functioning at day 45 | Day 45
  Improvement of GAF (Global Assessment of Functioning) scale between baseline and day 45
Evaluate the effect of tDCS on social adjustment at day 14 | Day 14
  Improvement of SAS (Social Adjustment Scale) scale between baseline and day 14
Evaluate the effect of tDCS on social adjustement at day 45 | Day 45
  Improvement of SAS (Social Adjustment Scale) scale between baseline and day 45

CONTACTS AND LOCATIONS:
Overall Officials: Nematollah JAAFARI, Professor, Study Director — Centre Hospitalier Henri Laborit
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: No